CLINICAL TRIAL: NCT00735774
Title: Suitability of 11C-ORM-13070 as a Positron Emission Tomography Tracer; an Open Study in Healthy Males
Brief Title: Suitability of 11C-ORM-13070 as a PET Tracer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Orion Corporation, Orion Pharma (Aila Holopainen, Clinical Study Director), Clinical study management
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 3099001
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Healthy volunteer study
MeSH Terms: interventions — 1-(1-(2,3-dihydrobenzo(1,4)dioxin-2-yl)methyl)-4-(3-methoxymethylpyridin-2-yl)piperazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 11C-ORM-13070 (Experimental)
  Interventions: Drug: 11C-ORM-13070

INTERVENTIONS:
Drug: 11C-ORM-13070 — Single dose of i.v. solution

SUMMARY:
The purpose of the study is to evaluate the suitability of 11C-ORM-13070 as a positron emission tomography tracer.

ELIGIBILITY:
Inclusion Criteria:

* Good general health ascertained by detailed medical history and physical examination
* Males between 18 and 45 years
* Body mass index (BMI) between 18-30 kg/m2
* Weight 55-95 kg (inclusive)

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastro-intestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator
* Any condition requiring regular concomitant medication including herbal products or likely to need any concomitant medication during the study.
* Regular consumption of more than 21 units of alcohol per week (1 unit = 4 cl spirits, about 13 g of alcohol)
* Current use of nicotine-containing products more than 5 cigarettes or equivalent/day
* Inability to refrain from using nicotine-containing products during the stay in the study centre
* Inability to refrain from consuming caffeine-containing beverages during the stay in the study centre e.g. propensity in getting headache when refraining from caffeine-containing beverages
* Blood donation or loss of significant amount of blood within 3 months prior to the screening visit
* Abnormal 12-lead electrocardiogram (ECG) finding of clinical relevance
* Any abnormal value of laboratory, vital signs, or physical examination, which may in the opinion of the investigator interfere with the interpretation of the test results or cause a health risk for the subject if he takes part into the study
* Anatomical abnormality in MRI which may in the opinion of the investigator interfere with the interpretation of PET results
* Participation in a drug study within 3 months prior to the entry into this study
* Participation in a prior PET study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Suitability of 11C-ORM-13070 as a PET tracer | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Juha Rinne, MD, PhD, Principal Investigator — Turku PET Centre
Locations (1):
- Turku PET centre, Turku, Finland